CLINICAL TRIAL: NCT01274845
Title: Use of Heliox in the Management of Neonates With Meconium Aspiration Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Tomasz Szczapa, Department of Neonatology at Poznań University of Medical Sciences
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 503-02-02215338-22961-03550
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Meconium Aspiration Syndrome
Keywords: Meconium aspiration syndrome; Heliox; Mechanical ventilation; Newborn
MeSH Terms: conditions — Meconium Aspiration Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heliox (Other)
  Interventions: Other: Heliox mechanical ventilation

INTERVENTIONS:
Other: Heliox mechanical ventilation — Mechanical ventilation (MV) with air-oxygen at baseline, then 1 hour of heliox (helium-oxygen) MV and then return to MV with air-oxygen.

SUMMARY:
The aim of the study: to assess the effect of short-term mechanical ventilation with heliox in newborns with meconium aspiration syndrome on vital signs, oxygenation, acid-base balance and respiratory function parameters.

ELIGIBILITY:
Inclusion Criteria:

* meconium aspiration syndrome diagnosed based on clinical and radiological findings,
* respiratory failure requiring mechanical ventilation

Exclusion Criteria:

* congenital malformations or congenital genetic syndromes,
* persistent pulmonary hypertension of the newborn (PPHN) requiring inhaled nitric oxide treatment

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Changes in acid-base balance and oxygenation | Parameters recorded first at the baseline during ventilation with air-oxygen gas mixture, then after 15 and 60 minutes of the heliox ventilation and finally 15 and 60 minutes after switching back to air-oxygen ventilation.
  Acid-base balance and oxygenation assessed on arterial blood gas samples, saturation measured with a pulse oximeter and calculated values of oxygenation index and alveolar-arterial oxygen tension difference.

SECONDARY OUTCOMES:
Changes in respiratory parameters | Parameters recorded first at baseline during ventilation with air-oxygen gas mixture, then after 15 and 60 minutes of the heliox ventilation and finally 15 and 60 minutes after switching back to air-oxygen ventilation.
  Analyzed parameters: tidal volume (VT, [ml/kg]), minute ventilation (VE, [l]) and peak expiratory flow rate (PEFR, [l/min]). Recorded ventilator settings: respiratory rate (RR), mean airway pressure (MAP) and fraction of inspired oxygen (FiO2).

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Szczapa, MD, PhD, Principal Investigator — Department of Neonatology at Poznań University of Medical Sciences
Locations (1):
- Department of Neonatology at Poznań University of Medical Sciences, Poznan, Poland